CLINICAL TRIAL: NCT06239194
Title: A Phase 1/2a, Multicenter, First-in-human, Open-label Clinical Trial Evaluating MDX2001 Monotherapy in Patients With Advanced Solid Tumors
Brief Title: Dose Escalation and Dose Expansion Study of MDX2001 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModeX Therapeutics, An OPKO Health Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MDX-2001-101
Record Dates: First submitted 2024-01-18; First posted 2024-02-02 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Biliary Tract Cancer; Breast Cancer; Cervical Cancer; Colon Cancer; Endometrial Cancer; Esophageal Cancer; Gastric Cancer; GastroEsophageal Cancer; Head and Neck Cancer; Hepatocellular Cancer; Non-small Cell Lung Cancer; Pancreatic Cancer; Prostate Cancer; Rectal Cancer; Renal Cancer; Thyroid Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Liver Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Prostatic Neoplasms; Rectal Neoplasms; Kidney Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 1a - MDX2001 Dose Escalation (Experimental): Patients with metastatic solid tumors will receive MDX2001 as intravenous (IV) infusion.
  Interventions: Drug: MDX2001
- Phase 1b - Dose Expansion - Dose A (Experimental): Patients with a single tumor indication receive MDX2001 as intravenous (IV) infusion.
  Interventions: Drug: MDX2001
- Phase 1b - Dose Expansion - Dose B (Experimental): Patients with a single tumor indication will receive MDX2001 as intravenous (IV) infusion.
  Interventions: Drug: MDX2001
- Phase 2a - Cohort Expansion (Experimental): Patients with a single tumor indication will receive MDX2001 as intravenous (IV) infusion at the recommended Phase 2 dose.
  Interventions: Drug: MDX2001

INTERVENTIONS:
Drug: MDX2001 — MDX2001 intravenous infusion

SUMMARY:
This study is designed to characterize the safety, tolerability, and anti-tumor activity of MDX2001 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study consists of Phase 1a dose escalation, Phase 1b dose expansion in a single indication, and Phase 2a expansion in a single indication.

Primary Objectives

* All Phases: Evaluate the safety and tolerability of MDX2001 in patients with advanced solid tumor malignancies
* Phase 1 only: Identify a recommended Phase 2 dose (RP2D) for further development of MDX2001
* For Phase 1b and Phase 2: Assess the anti-tumor efficacy of MDX2001 in patients with selected advanced solid tumor malignancies

Secondary Objectives:

* Further characterize the anti-tumor activity of MDX2001 based on additional assessments of clinical benefit
* Characterize the pharmacokinetics of MDX2001
* Characterize the immunogenicity of MDX2001
* Characterize relationship of baseline target protein expression in tumor tissue and clinical benefit

The expected duration of study intervention for patients may vary, based on progression date. The median expected duration of study per patient is estimated to be 10 months (up to 1 month for screening, a median of 6 months for treatment, and a median of 3 months for long term follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age
* Histologically or cytologically confirmed diagnosis of metastatic solid tumors
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* All patients should have at least 1 measurable disease per RECIST v1.1. An irradiated lesion can be considered measurable only if progression has been demonstrated on the irradiated lesion.
* All contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Adequate hematologic, hepatic and renal function
* Capable of giving signed informed consent

Exclusion Criteria:

* Any clinically significant cardiac disease
* Unresolved toxicities from previous anticancer therapy
* Prior solid organ or hematologic transplant
* Known untreated, active, or uncontrolled brain metastases
* Known positivity with human immunodeficiency virus (HIV), known active hepatitis B or C, or uncontrolled chronic or ongoing infectious requiring intravenous treatment.
* Receipt of a live-virus vaccination within 28 days of planned treatment start
* Patient not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions.
* Participation in a concurrent clinical study in the treatment period.
* Known hypersensitivity to MDX2001 or any of its ingredients

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
All Phases: Adverse events (AEs) | Baseline until end of study, up to approximately 9 months
  Incidence and severity of AEs and serious AEs (SAEs) graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 including changes in clinical laboratory parameters
Phase 1b and Phase 2a: Objective response rate of MDX2001 | From date of enrollment until the end of treatment, up to approximately 6 months
  Objective response rate is defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Phase 1: Recommended Phase 2 dose (RP2D) | Baseline until end of study, up to approximately 9 months
  Recommended Phase 2 dose is determined following the evaluation of MDX2001 safety including the incidences of dose limiting toxicities (DLTs), MDX2001 anti-tumor activity, and MDX2001 pharmacokinetics

SECONDARY OUTCOMES:
Phase 1a: Objective response rate of MDX2001 | From date of enrollment until the end of treatment, up to approximately 6 months
  Objective response rate is defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) per RECIST v1.1.
All Phases: Duration of response (DOR) | From date of enrollment until the end of treatment, up to approximately 6 months
  Duration of response is defined as the time from first documentation of response (complete response [CR] or partial response [PR]) to documentation of objective disease progression or death due to any cause, whichever occurs first
All Phases: Time to response (TTR) | From date of enrollment until the first documentation of response (CR or PR), approximately 4 months
  Time to response is defined as the time from first dose to first documentation of response (CR or PR)
All Phases: Disease control rate (DCR) | From date of enrollment until the end of treatment, up to approximately 6 months
  Disease control rate is defined as the proportion of evaluable patients with a best overall response (BOR) of stable disease, CR or PR
All Phases: Progression free survival (PFS) | From date of enrollment until the end of treatment, up to approximately 6 months
  Progression-free survival is defined as the time from the first dose to the date of disease progression or death (any cause), whichever occurs first
All Phases: Pharmacokinetic Parameter Cmax of MDX2001 | From date of enrollment until completion of the 6th cycle of treatment, up to approximately 6 months
  Maximum observed plasma concentration
All Phases: Pharmacokinetic parameter area under the curve (AUC(0-T)) of MDX2001 | From date of enrollment until the completion of the 3rd cycle of treatment, up to approximately 3 months
  Area under the plasma concentration versus time curve
All Phases: Evaluation of MDX2001 immunogenicity | Baseline until end of study, up to approximately 9 months
  The presence and persistence of anti-MDX2001 antibodies
All Phases: Correlation between tumor antigen expression and anti-tumor activity of MDX2001 | Baseline until the end of treatment, up to approximately 6 months
  Relationship between H score cell surface target protein expression in tumor tissue at baseline and objective responses with MDX2001

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Sarah Cannon Research Institute, Denver, Colorado
  - Sylvester Comprehensive Cancer Center - University of Miami Health System, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dumbrava E, Minchom A, Henry J, Johnson M, Sommerhalder D, Merchan J, Heist R, Cabanas EG, Cotreau M, Goenaga AL, Burzyn D, Makris L, Culm K, Abbadessa G. MDX-2001-101 study protocol: a phase I/IIa, multicenter, first-in-human, open-label clinical trial evaluating MDX2001 monotherapy in patients with advanced solid tumors. Future Oncol. 2026 Feb;22(3):305-312. doi: 10.1080/14796694.2025.2610468. Epub 2026 Jan 6. PMID 41495607